CLINICAL TRIAL: NCT05248659
Title: A Phase 2/3, Multicenter, Open-label Trial to Evaluate the Long-term Safety, Tolerability, and Efficacy of Sibeprenlimab Administered Subcutaneously in Subjects With Immunoglobulin A Nephropathy.
Brief Title: Phase 2/3 Open-Label Trial of Sibeprenlimab in the Treatment of Immunoglobulin A Nephropathy
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 417-201-00012
Record Dates: First submitted 2022-02-18; First posted 2022-02-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: Sibeprenlimab; VIS649; IgAN
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sibeprenlimab 400 mg s.c. q 4 weeks (Experimental)
  Interventions: Drug: Sibeprenlimab 400 mg s.c. Q4weeks

INTERVENTIONS:
Drug: Sibeprenlimab 400 mg s.c. Q4weeks — Sibeprenlimab 400 mg s.c. q 4 weeks
  Other Names: VIS649

SUMMARY:
This is a phase 2/3 open-label trial to evaluate the long-term safety, tolerability, and efficacy of sibeprenlimab administered subcutaneously (SC) in subjects with IgAN.

DETAILED DESCRIPTION:
This is a phase 2/3, multicenter, open-label trial to evaluate the long-term safety, tolerability, and efficacy of sibeprenlimab administered subcutaneously (SC) to subjects with IgAN.

Eligible subjects will have participated in trials 417-201-00007 or VIS649-201 and, in the investigator's judgement, could benefit from continued treatment with sibeprenlimab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed Trial 417-201-00007 or VIS649-201 without safety concerns and who, in the opinion of the investigator, could potentially benefit from treatment with sibeprenlimab.
* eGFR ≥ 20 mL/min/1.73 m2, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Exclusion Criteria:

* Subjects who have not completed participation in trials 417-201-00007 or VIS649-201.
* Subjects who, following enrollment in trials 417-201-00007 or VIS649-201 developed a condition or characteristic that would have excluded them from participation in these trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2028-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From baseline to the end-of-trial visit in Week 112.

SECONDARY OUTCOMES:
Annualized slope of Estimated Glomerular Filtration Rate (eGFR) | Over 12 and 24 months
Urine protein/creatinine ratio (uPCR) in a 24-hour collection | At 12 and 24 months
Proportion of Subjects with Clinical Remission as defined in the protocol | At 12 and 24 months
Time to Progression of Chronic Kidney Disease, as defined in the protocol | Over 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com